CLINICAL TRIAL: NCT01535755
Title: A Protocol to Wean From Noninvasive Mechanical Ventilation
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Enough patients has been enrolled.
Sponsor: Duan jun (Other)
Responsible Party: Sponsor-Investigator, Duan jun, The first affiliated hospital of chong qing medical univercity, Chongqing Medical University
Organization: Chongqing Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: cqykdxfsdyyy2
Record Dates: First submitted 2012-02-11; First posted 2012-02-20 (Estimated); Last update posted 2013-07-16 (Estimated); Status verified 2013-07

CONDITIONS: Ventilator Weaning
Keywords: noninvasive mechanical ventilation; ventilator weaning
MeSH Terms: interventions — Clinical Protocols

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- protocol group (Active Comparator): This group patients are weaned as the protocol which the investigators described.
  Interventions: Device: protocol
- clinicians' order group (Other): This group patients are weaned as the clinicians' order.
  Interventions: Other: physician's orders

INTERVENTIONS:
Device: protocol — In this group, the patients were weaned as the protocol.
  Other Names: In this group, the patients were weaned as the protocol.
  Arms: protocol group
Other: physician's orders — In this group, the patients were weaned as the clinicians' order.
  Other Names: In this group, the patients were weaned as the clinicians' order.
  Arms: clinicians' order group

SUMMARY:
The investigators use a protocol to wean from noninvasive mechanical ventilation.

DETAILED DESCRIPTION:
Design: Prospective, randomized, controlled trial, with 2 groups: study (protocol weaning group) and control (clinicians' order weaning group). Setting: Respiratory Intensive Care Unit (RICU). Subjects: Patients >18 yr, noninvasive mechanical ventilation >24 hours. Interventions and measurements: Study group (weaning as the protocol) and control group (weaning as the clinicians' order); recording of clinical variables at admission and during RICU stay, and end-point variables (noninvasive mechanical ventilation day, RICU and hospital stay, RICU mortality. Expected results: the protocol group's noninvasive mechanical ventilation days is less than clinicians' order group.

ELIGIBILITY:
Inclusion Criteria:

1. noninvasive mechanical ventilation > 24 hours.
2. age >18 years

Exclusion Criteria:

1. severe cerebraI，heart，hepatic and renal faiIure.
2. facial or cranial trauma or surgery.
3. facial abnormalities.
4. recent gastric or esophageal surgery.
5. active upper gastrointestinal bleeding.
6. large amount of sputum with weak cough ability
7. lack of co-operation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2010-07; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
The duration of noninvasive mechanical ventilation | from admission to ICU to discharge from it (average of 4 weeks)
  The duration of noninvasive mechanical ventilation was measured from the patients admitted to ICU to discharged from it,an expected average of 4 weeks.

SECONDARY OUTCOMES:
The successful weaning rate | from admission to ICU to discharge from it (average of 4 weeks)
  The successful weaning rate was measured from the patients admitted to ICU to discharged from it, an expected average of 4 weeks.
The length of ICU days | from admission to ICU to discharge from it (average of 4 weeks)
  The length of ICU days was measured from the patients admitted to ICU to discharged from it, an expected average of 4 weeks.
The intubation rate during the study | from admission to ICU to discharge from it (average of 4 weeks)
  The intubation rate during the study was measured from the patients admitted to ICU to discharged from it, an expected average of 4 weeks.
The mortality during the study | from admission to ICU to discharge from it (average of 4 weeks)
  The mortality during the study was measured from the patients admitted to ICU to discharged from it, an expected average of 4 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Jun Duan, Principal Investigator — The first affiliated hospital, Chongqing medical hospital
Locations (1):
- The first affiated hospital, chongqing medical university, Chongqing, Chongqing Municipality, China